CLINICAL TRIAL: NCT00223002
Title: Chlorhexidine Versus Povidone-Iodine for Prevention of Epidural Needle Contamination in the Parturient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BMC# 03-1315
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Asepsis; Analgesia, Epidural; Anesthesia, Epidural
MeSH Terms: conditions — Agnosia | interventions — Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): PI
  Interventions: Drug: Chlorhexidine
- 2 (Experimental): Chlorohex
  Interventions: Drug: Chlorhexidine

INTERVENTIONS:
Drug: Chlorhexidine — sample collected at time of procedure and then analysed for bacterial contamination

SUMMARY:
Infection after epidural catheter placement is fortunately rare. When it does happen, the affected person can become seriously ill.

This study examines which skin disinfectant, chlorhexidine or povidone-iodine, decreases the number of bacteria that can be grown from the skin washed with each disinfectant prior to placing an epidural catheter for pain control in labour.

DETAILED DESCRIPTION:
The use of chlorhexidine for skin asepsis for the placement of intravascular catheters is known to decrease the incidence of central line colonization and blood stream infection when compared to the use of povidone-iodine. While the development of an infectious complication following spinal or epidural analgesia, such as epidural abscess or meningitis, is fortunately rare, when it does happen, there can be devastating consequences for the affected individual. The low frequency of infection makes a trial with an endpoint of clinical infection not feasible, however a reduction in skin and needle contamination following attempts at asepsis should reduce the risk of infectious complication. Ongoing work by the authors is examining the skin culture rates following randomized standardized skin disinfection. The purpose of this randomized trial is to compare needle culture rates to further assess effectiveness of skin disinfection following a standardized skin preparation with either povidone-iodine or chlorhexidine in pregnant women requesting lumbar epidural pain relief in labour.

ELIGIBILITY:
Inclusion Criteria:

* Parturients requesting lumbar labour epidural analgesia while investigator is assigned to the Obstetrical Anesthesia Service

Exclusion Criteria:

* Known allergy to either skin disinfectant
* Requirement to receive antibiotics prior to placement of lumbar epidural catheter
* Immunosuppression of the participant

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2004-11; Primary Completion 2007-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
culture-positive rate of epidural needles processed by microbiology lab | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Susan A Shaw, MD, Principal Investigator — University of Saskatchewan College of Medicine
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada